CLINICAL TRIAL: NCT06597487
Title: Influence of Wolters Classification of Pulpitis and the Radiographic Caries Depth Detected Using Artificial Intelligence on the Success of Full Pulpotomy in Permanent Mature Molars With Irreversible Pulpitis: A Randomized Controlled Trial
Brief Title: The Effect of Prognostic Factors on the Success of Full Pulpotomy in Permanent Mature Molars With Irreversible Pulpitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Principal Investigator, Mayand Amer Mohamed Yehia Amer, Principal Investigator, Misr International University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MIU-IRB-2324-039
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Pulpitis - Irreversible
Keywords: irreversible pulpitis; full pulpotomy; artificial intelligence

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Root Canal Treatment (Active Comparator): The patients allocated to this arm will receive conventional root canal treatment. They will be followed up for 1, 3 and 6 months to assess clinical and radiographic success.
  Interventions: Procedure: Conventional root canal treatment
- Full Pulpotomy (Experimental): The patients allocated to this arm will receive full pulpotomy. They will be followed up for 1, 3 and 6 months to assess clinical and radiographic success.
  Interventions: Procedure: Full pulpotomy

INTERVENTIONS:
Procedure: Full pulpotomy — The patients will receive full pulpotomy as follows:
  -Under rubber dam isolation, the operator will perform caries removal, complete the access cavity preparation, achieve hemostasis from all canals, and apply the bioceramic material. The operator will seal the cavity with glass ionomer restoration.
  Arms: Full Pulpotomy
Procedure: Conventional root canal treatment — The patients will receive conventional root canal treatment, which is the gold standard treatment protocol in cases with irreversible pulpitis.
  Arms: Root Canal Treatment

SUMMARY:
This study aims to evaluate the effect of prognostic factors, such as the degree of pulpal inflammation and the radiographic caries depth, on the success of full pulpotomy in mature permanent molars with irreversible pulpitis.

DETAILED DESCRIPTION:
* Patients with mature permanent molars diagnosed with irreversible pulpitis will be enrolled in the study.
* The pre-operative pulpal status will be assessed using the American Association of Endodontists (AAE) classification and Wolters classification.
* Pre-operative radiographs will be taken, and radiographic caries depth will be assessed.
* An Artificial Intelligence software will process the pre-operative X-rays to assess the presence of carious pulp exposure. The diagnostic accuracy of the software will be evaluated by comparing its readings with clinical findings of pulp exposure after caries removal.
* The patients will be randomized to receive either full pulpotomy or conventional root canal treatment.
* The patients will be followed up for 1, 3 and 6 months to assess clinical and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

* Mature permanent molars with irreversible pulpitis.
* Presence of bleeding pulp tissues from all canals.
* The tooth is not periodontally compromised.

Exclusion Criteria:

* Non-vital teeth.
* Uncontrolled bleeding from any of the canals after ten minutes of application of hemostatic agent.
* Molars with immature roots.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Percentage of Successful Cases | After 1, 3, and 6 months
  * It will be measured as a percentage.
  * It will be decided according to the clinical and radiographic criteria of success and failure.
Diagnostic accuracy (Sensitivity and Specificity) of an artificial intelligence software in detecting carious pulp exposure | On the day of the procedure
  * The Artificial Intelligence (AI) software will process pre-operative radiographs to predict the presence of carious pulp exposure. The AI findings will be compared to the clinical findings of carious pulp exposure after caries removal. (Clinical finding of carious pulp exposure will be used as the gold standard).
  * The outcome will be reported as Sensitivity and Specificity.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Ghobashy, Prof. Dr., Study Director — Misr International University
Locations (1):
- Misr International University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided